CLINICAL TRIAL: NCT00000238
Title: Temporal Discounting Delayed Outcomes on Opioid-Dependent Outpatients
Brief Title: Temporal Discounting Delayed Outcomes on Opioid-Dependent Outpatients - 20
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Purpose: Treatment
Other Study IDs: NIDA-06969-20; R01-06969-20
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to assess the degree in which opioid-dependent outpatients discount the value of an additional maintenance dose of buprenorphine under differing states of opioid deprivation.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-08

PRIMARY OUTCOMES:
Drug use
Money choice
Heroin craving

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States